CLINICAL TRIAL: NCT03510819
Title: Evaluation of Knowledge- Attitude- Practice (KAP) of Intern Dentists in Emergency Management of Traumatic Dental Injuries in Permanent Anterior Teeth: A Cross-sectional Study
Brief Title: Evaluation of Knowledge- Attitude- Practice (KAP) of Intern Dentists in Emergency Management of Traumatic Dental Injuries in Permanent Anterior Teeth
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Nada Mahmoud Shaheen, B.D.S 2013, Cairo University
Other Study IDs: CEBD-CU-2018-04-11
Record Dates: First submitted 2018-04-10; First posted 2018-04-27 (Actual); Last update posted 2018-04-27 (Actual); Status verified 2018-04

CONDITIONS: Traumatized Permanent Anterior Teeth
Keywords: Dental trauma; Emergency management; Tooth avulsion; Knowledge; Practice; Traumatic injuries; Attitude
MeSH Terms: conditions — Tooth Avulsion; Wounds and Injuries; Behavior

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This study aims to evaluate knowledge, Attitude and Practice of intern dentists in emergency management of traumatic dental injuries in permanent anterior teeth in children aged from 6 to 12 years old. A questionnaire survey will be designed to evaluate Knowledge - Attitude - and practice (KAP) of intern dentists who met the eligibility criteria.

ELIGIBILITY:
Inclusion Criteria:

* Intern dentists attending their internship in Faculty of Dentistry- Cairo University, other private university (Modern Science and Arts University- MSA).
* The intern dentists who agree to participate.
* Intern dentists who did not attend Pediatric Dentistry round, Endodontic round, Emergency round and Surgery round at Cairo University.
* Intern dentists irrespective of age and sex.

Ages: 22 Years to 23 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Dentists attending their internship in Cairo University and another private university (Modern Science and Arts University- MSA).
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2018-04-01 (Actual); Primary Completion 2019-04-15 (Estimated); Study Completion 2019-05-15 (Estimated)

PRIMARY OUTCOMES:
Knowledge, attitude and practice (KAP) of intern dentists. | 1 year
  Measured by a KAP questionnaire and the measuring Unit is Binary ( Yes, No)
Knowledge, attitude and practice (KAP) of intern dentists. | 1 year
  Measured by a KAP questionnaire and the measuring Unit is Multiple choice questions.

CONTACTS AND LOCATIONS:
Locations (1):
- Cairo University, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Undecided